CLINICAL TRIAL: NCT05914844
Title: The Role Of Hyaluronan Receptor Cd44s And Has2 In Endometrial Malignities
Brief Title: Investigation Of Receptivity Markers For Endometrial Cancer Treatment Development
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Hayrunnisa Yesil Sarsmaz, Asistant Prof., Celal Bayar University
Other Study IDs: MCBU_endometriumcancer
Record Dates: First submitted 2022-12-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Endometrial Cancer Stage
Keywords: endometrial carcinoma; immunohistochemistry; CD44s; HAS2
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial tissue cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1:: Proliferative phase endometrium (PPE)
- Group 2:: Secretory phase endometrium
- Group 3:: Benign endometrial hyperplasia
- Group 4:: Endometrial intraepithelial neoplasia
- Group 5:: Early stage of endometrial carcinoma
- Group6:: Advanced stage of endometrial carcinoma

SUMMARY:
Hyaluronan is an extracellular matrix protein that is involved in cell-cell and cell-matrix interactions. Hyaluronan performs this activity through hyaladherins, which are intracellular and extracellular receptors.

The purpose of this study was to compare the distributions of Hyaluronan Synthetase 2 (HAS2) and CD44s in healthy endometrial tissue samples obtained during the proliferative phase endometrium (PPE) and secretory phase endometrium (SPE), as well as pathologic samples diagnosed with benign endometrial hyperplasia (EH), endometrial intraepithelial neoplasia (EIN), early stage of endometrial carcinoma (EC) (stage I/II) and advanced stage of endometrial carcinoma (stage III/IV) (n:5, each).

By using the avidin-biotin-peroxidase method, tissue samples that had been fixed with formalin passed through a regular paraffin follow-up protocol, and subsequently embedded in paraffin were stained indirectly with anti-CD44s and anti-HAS2 primary antibodies. Immunostaining intensity was graded as 0: negative, 1: weak, 2: moderate, 3: strong, and 4: very strong using a semiquantitative technique. The ANOVA test was used to assess the statistical significance of the findings. Statistical significance was defined as (p) values less than 0.05.

While weak HAS2 and weak/moderate CD44s immunoreactivity was observed on the surface epithelium (SE)/glandular epithelium (GE) and stroma of the tissue samples acquired during PPE; weak/moderate HAS2 and moderate CD44s immunoreactivity were observed in SPE and EH groups; moderate/strong HAS2, strong CD44s immunoreactivity was observed in EIN; strong/very strong HAS2 and very strong CD44s immunoreactivity were observed in early-stage EC and advanced stage EC. It was determined that the immunoreactivity intensity increased at a statistically significant level in both early and advanced stage EC.

The fact that HAS2 and CD44s, two intracellular receptors, have increased in endometrial carcinoma leads us to believe that they are likely to play a role in tumor development, invasion, migration, metastasis and that they may be useful in developing future treatment protocols targeting hyaluronan receptors.

ELIGIBILITY:
Inclusion Criteria:

- All patients with endometrial carcinoma underwent surgery.

Exclusion Criteria:

* No patient was subject to chemotherapy or radiotherapy prior to surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with endometrium cancer
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Investigation Of Receptivity Markers For Endometrial Cancer Treatment Development | Baseline
  The increase or decrease of hyaluronan receptors, which play a role in endometrial cancer, has a critical role to be explained in cancer treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Yunusemre, Mani̇sa, Turkey (Türkiye)